CLINICAL TRIAL: NCT05228522
Title: Preventing Diabetes in Latino Families
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: St. Vincent de Paul Medical and Dental Clinic (Other); Valley of the Sun YMCA, Arizona (Other); University of Washington (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DK107579-06A1 (NIH); 1R01DK107579-01 (NIH)
Record Dates: First submitted 2022-01-05; First posted 2022-02-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes; Obesity; Pediatric Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Intervention (Experimental): 16-week family-focused intervention that includes nutrition education, behavioral change skills training, and physical activity.
  Interventions: Behavioral: Lifestyle Intervention
- Comparison control (No Intervention): Comparison control families meet with the Study Physician and a Registered Dietitian as a family to review laboratory results and receive lifestyle counseling. Control families will be contacted on a monthly basis for a total of 12 months.

INTERVENTIONS:
Behavioral: Lifestyle Intervention — 16-week family-focused intervention that includes nutrition education, behavioral change skills training, and physical activity.
  Arms: Lifestyle Intervention

SUMMARY:
Purpose: This study will test the efficacy of a family-focused lifestyle intervention for reducing type 2 diabetes (T2D) risk factors and increasing Quality of Life (QoL) among high-risk Latino families.

DETAILED DESCRIPTION:
Background: T2D disproportionately impacts Latino children, families and communities. The Diabetes Prevention Program (DPP) established that T2D can be prevented in high-risk adults through intensive lifestyle intervention. Although the DPP has been translated to a variety of adult populations and settings, engagement and effectiveness is diminished in minority communities and there are no family-focused diabetes prevention trials for Latinos. The culturally-grounded approach is guided by an Ecodevelopmental model that considers community, family, peer, and individual-level factors that influence health behaviors and health outcomes over time. The study will test the efficacy of a 16-week family-focused lifestyle intervention for reducing T2D risk and increasing QoL among high-risk Latino families as compared to control families. The study will use Integrative Mixed Methods to understand how family structures and processes influence intervention outcomes.

ELIGIBILITY:
Inclusion/Exclusion Criteria - Children

Inclusion

* Latino: self-report
* Age: 10-16 years
* Obesity: BMI ≥ 95th percentile for age and sex

Exclusion

* Type 2 diabetes: (standard American Diabetes Association criteria)
* Taking medication(s) or diagnosed with a condition that influences carbohydrate metabolism, physical activity, and/or cognition
* Currently enrolled in (or within previous 12 months) a formal diabetes prevention or weight loss program
* Self-identify as American Indian
* Unstable depression or other mental health condition that may impact QoL

II. Inclusion/Exclusion Criteria - Parents

Inclusion

• Parent of a child who meets the above child inclusion/exclusion criteria

Exclusion

* Currently enrolled in (or within previous 12 months) a formal diabetes prevention or weight loss program
* Self-identify as American Indian

Ages: 10 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-12-12 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Glucose Tolerance | 16 weeks
  Glucose tolerance will be determined using a standard 75-gram Oral Glucose Tolerance Test (OGTT) with samples collected at fasting and 120 minutes for assessment of glucose concentrations. We will follow the OGTT protocol used by the CDC for the NHANES.
  Centers for Disease Control. Oral Glucose Tolerance Test (OGTT) Procedures Manual. In: Survey NHaNE, ed2007.

SECONDARY OUTCOMES:
Weight Specific Quality of Life (QoL) | 16 weeks
  Youth Quality of Life (YQOL) inventory shows strong psychometric properties, internal consistency (Chronbach's alpha >0.80), test-retest reliability (ICC > 0.74), and construct validity with other pediatric QoL measures (r = 0.73, P<0.05 with KINDL).
  Weight-specific QoL (YQOL-W) measures three domains of weight-related QoL (Self, Social, Environmental). The instrument shows good reliability (ICC = 0.77) and construct validity with the Children's Depression Inventory (r=0.57, P<0.01).
  Adults will be assessed using the World Health Organization Brief Quality of Life Instrument, demonstrates good to excellent psychometric properties. Weight-specific QoL in adults will be assessed by the Obesity and Weight-Loss Quality of Life (OWLQOL) instrument which demonstrates strong psychometric properties internal consistency (Chronbach's alpha >0.90), test-retest reliability (ICC > 0.95), and construct validity with other QoL measures (r = 0.53, P<0.05).
Total body composition-muscle | 16 weeks
  Muscle (grams) will be assessed by Dual-energy X-Ray Absorptiometry (DXA) using the GE Lunar iDXA (GE Lunar, Madison, WI).
Total body composition-fat | 16 weeks
  Fat (grams) will be assessed by Dual-energy X-Ray Absorptiometry (DXA) using the GE Lunar iDXA (GE Lunar, Madison, WI).
Total body composition-bone | 16 weeks
  Bone density (grams) will be assessed by Dual-energy X-Ray Absorptiometry (DXA) using the GE Lunar iDXA (GE Lunar, Madison, WI).
Physical Activity | 16 weeks
  Physical Activity will be assessed using accelerometers (Actigraph wGT3X-BT) to capture minutes/day of moderate, moderate to vigorous, and vigorous activity over 7-days with >4 days and >10 hours/day determined as valid. Data will be processed and analyzed using ActiLife v6.13 software.
Dietary behaviors | 16 weeks
  Dietary behaviors will be assessed using the NCI ((National Cancer Institute) Dietary Screener Questionnaire.
  To score the questionnaire, we use the NCI's (National Cancer Institute) scoring algorithms to convert screener responses to estimates of individual dietary intake for fruits and vegetables (cup equivalents), dairy (cup equivalents), added sugars (teaspoon equivalents), whole grains (ounce equivalents), fiber (g), and calcium (mg) with higher values indicating greater intake. For a fuller description of the statistical methods used, see: Thompson FE, Midthune D, Kahle L, Dodd KW. Development and Evaluation of the National Cancer Institute's Dietary Screener Questionnaire Scoring Algorithms. J Nutrition 2017 Jun;147(6):1226-1233.

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
We will share aggregate data but no individual participant data will be shared with other researchers.